CLINICAL TRIAL: NCT05998577
Title: A Personalized Approach to Abdominal Pain in Irritable Bowel Syndrome and Inflammatory Bowel Disease Using Experience Sampling Method (ESM) and a Digital Food Diary (Traqq)
Brief Title: A Personalized Approach to Abdominal Pain in Irritable Bowel Syndrome
Acronym: PERCEPTIvE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL82286.068.22
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Irritable Bowel Syndrome; Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Functional Gastrointestinal Disorders; Lifestyle Factors
Keywords: Experience Sampling Method; Traqq
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESM/Traqq (Experimental): Use of ESM and Traqq for one week to get a personalised analysis of the abdominal pain and triggerfactors that can be used at the outpatient clinic visit to select an effective treatment option.
  Interventions: Device: ESM and Traqq
- Standard care (No Intervention): Will not be using ESM and Traqq, but will only get a standard outpatient clinic visit together with PDSkeuzehulp to make a decision for a treatment.

INTERVENTIONS:
Device: ESM and Traqq — Two telephone applications: ESM is a psychosocial diary and Traqq is a food diary to measure abdominal pain as well as possible triggerfactors (i.e. diet, stress, anxiety)
  Arms: ESM/Traqq

SUMMARY:
Apart from its use to provide insight in IBS disease courses and in clinical research, ESM can provide patients with feedback about individual triggers of their symptoms, and thereby function as part of a personalized therapeutic strategy. This is also true for IBD-IBS. Treatment strategies in IBS and IBD-IBS are largely based on reassurance, identification and elimination of triggering factors, and in more severe cases pharmaco- and psychotherapy. The ESM approach has the potential to increase therapeutic efficacy in IBS and IBD-IBS and will assist patients in disease self-management. The Traqq application can provide more detailed information about the dietary pattern of IBS and IBD-IBS patients. Traqq in combination with ESM will give an overview of abdominal pain and associated symptoms and psychosocial factors are exposed to during the day. The insight provided using ESM and Traqq may improve patient understanding of their personal symptom dynamics and triggers, as well as the physician's insight into the symptom patters of the specific patients, which may aid treatment choice and eventually improve the outcome of any treatment provided in daily clinical care.

DETAILED DESCRIPTION:
This is an unicenter, prospective, proof-of-concept randomized controlled, non-blinded intervention study that focuses on two patient populations, with overlapping symptom patterns and treatment approaches, i.e. patients with IBS and IBD-IBS.

Following written informed consent, the eligibility screening is performed and instructions about the study procedures will be given. Hereafter, both groups will independently be randomized into i) an ESM/Traqq arm or ii) a standard care arm. The intervention group and the control group will complete the IBS-SSS, EO-5D-5L, GAD-7, PHQ-9, VSI, and MFl-20 as well as the Rome IV criteria for IBS and functional dyspepsia at baseline and the intervention group will complete thereafter the ESM and Traqq applications during the first week. After this week, the data will be analysed to identify associations between abdominal pain and psychosocial factors, diet or other GI associated symptoms. About two weeks later, participants will have their second visitation at the outpatient clinic with their treating physician. In the intervention group, but not the control group, the patient and the treating physician will receive the results of the personal data of the patients based on ESM and Traqq. The insight participants and their physicians get from this information, will help them to make changes in lifestyle factors that affect their symptoms or to choose a pharmacological or non-pharmacological treatment. However, the study protocol will not indicate which treatment choice should be made by the patient and their treating physicians. That choice will still be based on shared decision making, just as in the standard care arm, only with the additional data provided. Furthermore, if the patients are referred to a dietician, psychologist, or both, the digital data obtained in the intervention group can be used to personalize the therapy. After giving informed consent by the participant for the data of ESM and Traqq being sent to the dietician or psychologist they are referred to, the coordinating investigator will send the data digitally to the dietician or psychologist that is needed for the personalized treatment. Participants in the control arm will get a consultation with the gastroenterologist as usual after the same period of time as the intervention group get their consultation. The participants of the control group will be given treatment advice only based on this consultation, the PDSkeuzehulp by shared decision making, according to standard care. Twelve weeks after the second outpatient visit, independently of the chosen treatment approach, the participants in both study groups will be asked to complete IBS-SSS, EQ-5D-5L, GAD-7, PHO-9, VSI, MFI-20 and Rome IV criteria for IBS and functional dyspepsia for the second time to evaluate whether there is an effect on 1) reduction of abdominal pain and 2) quality of life, psychological aspects or fatigue of the participants due to the insight provided by ESM and Traqq.

After those twelve weeks, the coordinating investigator will contact the participants of the intervention group and control group by phone for the last time. Participants are asked what treatment they have gotten and what lifestyle modifications they have done to reduce abdominal pain. To improve compliance for completing the questionnaires by the control group, the participants in the control group will get the opportunity to use the ESM and Traqq applications after the study has been completed. This will not be part of this study but can be beneficial for those individuals who have not got any additional insight about their symptoms by getting the standard care.

ELIGIBILITY:
Inclusion criteria IBS patients

* A diagnosis of IBS according to Rome IV criteria, as follows:

  * Recurrent abdominal pain, on average, at least 1 day per week in the last 3 months, associated with 2 or more of the following criteria:
  * Related to defecation;
  * Associated with a change in stool frequency; oAssociated with a change in stool form (appearance).
  * Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.
* Minimal baseline score of 150 points on the IBS-SSS scale
* Age between 18 and 70 years;
* Ability to understand and speak the Dutch language
* Ability to understand how to utilize the ESM and Traqq applications.

Inclusion criteria IBD patients

* Patients with IBD diagnosed in accordance with current ECCO guidelines, with IBD- IBS and with chronic abdominal pain, as follows:

  * MIAH score <3
  * Fecal calprotectin < 150 ug/g
  * Fulfilling the Rome IV criteria for IBS.
* Age between 18 and 70 years;
* Minimal baseline score of 150 points on the IBS-SSS scale
* Ability to understand and speak the Dutch language
* Ability to understand how to utilize the ESM and Traqq applications.

Exclusion criteria IBS patients

* Any organic explanation for the abdominal symptoms;
* A history of abdominal surgery, except for uncomplicated appendectomy, laparoscopic cholecystectomy and hysterectomy is present;
* Pregnant or lactating at the baseline visit.

Exclusion criteria IBD patients

* Uncertainty about the absence of active inflammation
* Uncertainty about other explanatory causes for the GI symptoms, such as bile acid malabsorption, intestinal stenosis, or small intestinal bacterial overgrowth;
* Pregnant or lactating at the baseline visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-05-19 (Estimated); Study Completion 2025-05-19 (Estimated)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome- Symptom Severity Score (IBS-SSS) | 12 weeks after outpatient clinic visit
  Change in IBS-SSS to see whether IBS symptoms are improved
  Scale 0-500 A higher score means worse outcome

SECONDARY OUTCOMES:
General Anxiety Disorder-7 (GAD-7) | 12 weeks after outpatient clinic visit
  Change in GAD-7 to see whether complaints of anxiety are improved
  Scale 0-21 A higher score means worse outcome
Multidimensional Fatigue Inventory-20 (MFI-20) | 12 weeks after outpatient clinic visit
  Change in MFI-20 to see whether fatigue is improved
  Scale 20-100 A higher score means worse outcome
Patient Health Questionnaire-9 (PHQ-9) | 12 weeks after outpatient clinic visit
  Change in PHQ-9 to see whether complaints of depression are improved
  Scale 0-27 A higher score means worse outcome
Visceral Sensitivity Index (VSI) | 12 weeks after outpatient clinic visit
  Change in VSI to see whether complaints of GI related anxiety are improved
  Scale 0-75 A higher score means worse outcome
European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) | 12 weeks after outpatient clinic visit
  Change in EQ-5D-5L to see whether quality of life is improved
  Scale 5-25 A higher score means worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All research data will be saved as an SPSS file with all available metadata such as variables, value labels and definitions of missing data in accordance with the existing codebooks. In addition, the research data will be saved as csv files. After completion of the study, the data will be archived and the data will be stored in accordance with the required format of the relevant data archive.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code